CLINICAL TRIAL: NCT04926701
Title: A First in Human Randomised, Double Blind, Placebo-controlled, Two-part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses (SAD and MAD) of Inhaled ETD001 in Healthy Male and Female Subjects
Brief Title: A First in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Inhaled ETD001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enterprise Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-ENAC-01
Record Dates: First submitted 2021-06-10; First posted 2021-06-15 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single ascending dose (Experimental): Single dose of inhaled ETD001/placebo on one occasion
  Interventions: Drug: ETD001 single dose; Drug: Placebo single dose
- Multiple ascending dose (7 days) (Experimental): Daily doses of ETD001/placebo for 7 consecutive days
  Interventions: Drug: ETD001 multiple twice daily doses; Drug: Placebo multiple twice daily doses; Drug: ETD001 multiple once daily doses; Drug: Placebo multiple once daily doses
- Multiple ascending dose (14 days) (Experimental): Daily doses of ETD001/placebo for 14 consecutive days
  Interventions: Drug: ETD001 multiple twice daily doses; Drug: Placebo multiple twice daily doses

INTERVENTIONS:
Drug: ETD001 single dose — Single ascending doses of inhaled ETD001
  Arms: Single ascending dose
Drug: Placebo single dose — Single doses of inhaled placebo
  Arms: Single ascending dose
Drug: ETD001 multiple twice daily doses — Ascending doses of inhaled ETD001 administered twice daily
  Arms: Multiple ascending dose (14 days); Multiple ascending dose (7 days)
Drug: Placebo multiple twice daily doses — Doses of inhaled placebo administered twice daily
  Arms: Multiple ascending dose (14 days); Multiple ascending dose (7 days)
Drug: ETD001 multiple once daily doses — Doses of inhaled ETD001 administered once daily
  Arms: Multiple ascending dose (7 days)
Drug: Placebo multiple once daily doses — Doses of inhaled placebo administered once daily
  Arms: Multiple ascending dose (7 days)

SUMMARY:
This is a first in human study of ETD001 a new drug being developed for the treatment of cystic fibrosis. The study is a randomised, placebo-controlled, double-blind interventional study to assess the safety, tolerability and pharmacokinetics of single and multiple ascending doses of inhaled ETD001in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females using suitable methods of contraception, or females of non-childbearing potential
* Consent to study participation
* Body weight ≥ 50 kg and body mass index 19 - 30 kg/m2
* Vital sign assessments within the normal ranges
* Healthy as determined following physical and laboratory examinations at screening visit
* Spirometry readings (FEV1 and FVC) to be ≥ 80% of predicted value

Exclusion Criteria:

* Acute or chronic illness detected at the screening visit
* Respiratory tract infection within 4 weeks of the screening visit
* Use of prescribed or OTC medication within 14 days of the screening visit
* History of regular alcohol use over the recommended limits within 6 months of screening, or history/evidence of alcohol or drug abuse
* Smoker or use of tobacco products within 6 months of screening
* Abnormal blood or urine laboratory test results at screening
* Recent participation (within 3 months) in another clinical trial
* Current, or history of, allergy that may be contraindicated

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting one or more treatment emergent adverse event (TEAE) | Baseline to Week 8
Number of participants who discontinue due to an adverse event (AE) | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for 12-lead ECG assessment at least once post dose | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for vital signs assessments at least once post dose | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for laboratory assessments at least once post dose | Baseline to Week 8
Number of participants who meet the markedly abnormal criteria for spirometry assessments at least once post dose | Baseline to Week 8

SECONDARY OUTCOMES:
Plasma concentrations of ETD001 | Day 1 pre-dose and at multiple time-points (up to 14 days) post final dose
  Blood levels of ETD001 measured after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Niyati Prasad, MD, Study Director — Enterprise Therapeutics
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom